CLINICAL TRIAL: NCT00265369
Title: Comparative Efficacy and Safety of a Bacillus Clausii Probiotic Strain Versus Placebo in the Treatment of Acute Diarrhoea in Children
Brief Title: TEDDY: Spores of Bacillus Clausii in Acute Diarrhoea in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C_9240
Record Dates: First submitted 2005-11-04; First posted 2005-12-14 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

INTERVENTIONS:
Drug: Spores of Bacillus Clausii Probiotic Strain

SUMMARY:
Primary objective:

* To demonstrate the efficacy of a Bacillus clausii probiotic strain compared to placebo in children suffering from acute diarrhoea and treated for 7 days.

Secondary objective:

* To evaluate the clinical safety of the Bacillus clausii probiotic strain versus placebo.

ELIGIBILITY:
Inclusion criteria:

Infants or Children

* Non hospitalized infants or children
* With acute diarrhea evident for less than 48 hours
* Having had three or more watery stools during the preceding 24 hours

Exclusion criteria:

Infants or Children

* With blood stools
* Having been treated with antibiotics or probiotics within the two weeks before the enrollment
* Suffering from dehydration defined by a weight loss of at least 5% or by the presence of a skin fold
* With an history of seizures
* With immunosuppressive conditions
* With a current status requiring an antibiotic treatment
* Suffering from a chronic disease including chronic diarrhea whatever the origin
* Having received before inclusion one of the following treatments:

  * Probiotics
  * Prebiotics
  * Drugs with adsorbing properties
  * Drugs that modify intestinal secretion like bismuth subsalicylate, acetorphan
  * Drugs that modify intestinal motility (opiates such as loperamide, atropine and other cholinergic agents).
* Having participated in another clinical trial in the last 3 months prior to the start of the study

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420
Dates: Start 2004-05

PRIMARY OUTCOMES:
Duration of diarrhoea as counted from the first intake of the investigational product up to the first appearance of a loose stool followed by two-consecutive normal stools

SECONDARY OUTCOMES:
Number of infants/children with normal stools at D3, D4, D5, D6 and D7;Mean number of stools per day;Occurrence of vomiting episodes per day after enrolment;Parents'overall global assessment of efficacy at the end of the treatment;other safety criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Perdriset, MD, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, Paris, France